CLINICAL TRIAL: NCT00164307
Title: Assisting Children With Prenatal Alcohol Exposure in Developing Peer Friendships
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: CDC-NCBDDD-3642; U84/CCU9201158-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2005-11-08 (Estimated); Status verified 2005-09

CONDITIONS: Treatment; Control

INTERVENTIONS:
Behavioral: Parent assisted social skills training

SUMMARY:
Children will be randomly assigned to a Parent-assisted social skills training or Wait list. Baseline and post intervention rating will be obtained from teachers.

DETAILED DESCRIPTION:
Targeted Area of Intervention: Social skills and development of best friend relationships. The specific intervention will be twelve small group sessions (90 minutes each) over a 6-week period. Child sessions consist of 4 components: 1) children report on homework assignments; 2) didactic presentation, behavioral rehearsal, and coaching, 3) coached play, and 4) new homework activities assigned with parent. Topics to be addressed across sessions include: reduction of maladaptive behaviors, information exchange techniques, places and times to make friends, group acceptance, praising other children, negotiation, play dates, dealing with teasing, and winner/loser skills. At the start of the intervention, parent and children will work with staff to develop a list of social skills, behaviors, and goals that they would like targeted for each child.

Parent component: Kathleen Mitchell (NOFAS) is an investigator to provide parent input to the study. Parent-only sessions will instruct them on key features being taught to their child. Concurrent parent sessions will include: 1) education on FAS/ARND, 2) parents present specific issues with their child, 3) review of current child session objectives and techniques, 4) new homework activities developed, 5) parent and child together review homework.

Evaluation Plan: Treatment and control (WL) groups will be compared using pre- and post-tests measures. Post-tests will be at the conclusion of the intervention and at a 4-month follow-up. Baseline parent measures include Social Skills Rating Scale, FAS Behavior Scale, and Test of Advocacy Knowledge. Baseline child measures include knowledge of social skills. Process (e.g., homework completion, attendance, etc) and outcome (e.g., social skills ratings, progress towards individual goals) measures will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* children ages 6 to 8 years
* history of prenatal alcohol exposure

Exclusion Criteria:

* non english speaking

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100
Dates: Start 2001-10; Study Completion 2005-01

PRIMARY OUTCOMES:
social skills
peer relationships/friendships

CONTACTS AND LOCATIONS:
Overall Officials: Mary O'Connor, PhD, Principal Investigator — University of Califorrnia at Los Angeles
Locations (1):
- University of California, Los Angeles, California, United States